CLINICAL TRIAL: NCT05541458
Title: Alleviating Chronic Morbidities and Food Insecurity by Launching a Food-as-medicine Program Called: The Good Food Rx
Brief Title: The Good Food Rx: Food-as-medicine Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency); Well Fed (Unknown); Arkansas Community Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 274352
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Diabetes Mellitus; Obesity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Obesity | interventions — Food; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Educational sessions plus a nutrition box and recipes (Experimental): Monthly nutrition education sessions will be attended by the subjects and then each subject will receive a free nutrition box that includes recipes that pertain to the food contents in the prepackaged box
  Interventions: Other: Food as medicine

INTERVENTIONS:
Other: Food as medicine — * Encourage participants to make dietary changes by increasing consumption of nutritious foods, particularly fruits and vegetables.
  * Reduce food insecurity by making it easier for participants to access nutritious foods to ensure they are eating a balanced diet.
  * Increase nutrition literacy.
  * Improve health-related outcomes of participants by decreasing chronic health conditions by decreasing health metrics using food as medicine.

SUMMARY:
This pilot study seeks to recruit 25 participants who meet program criteria by alleviating chronic morbidities that plague this region by providing participants with nutritional food boxes partnered with nutrition education classes to determine impact and potential benefits of using food as medicine. The key measures seeking to be examined in the program are reducing food insecurity, healthy food consumption, increased nutrition education, and a decrease in biometrics such as hypertension, A1C levels, hyperlipidemia indices, and obesity.

UAMS East seeks to alleviate chronic morbidities and food insecurity by launching a food-as-medicine program called The Good Food Rx. The Good Food Rx Program couples established nutrition education classes participation with, at the same time, providing healthy curated nutritional food boxes to at-risk individuals.

DETAILED DESCRIPTION:
Study Design and Procedures In this study, the Principal Investigator, Director of Outreach, Food RX Program Coordinator and/or Heath Educator are considered "study personnel."

The chronological study design of The Good Food Rx program are as follow:

* Participants will be identified for study/program participation by the Principal Investigator using medical health records and/or a referral from a UAMS East nurse or doctor. Flyers will also be present in the clinic for participant attraction. Prospective participants inquiring about the study will have their medical records reviewed by the Principal Investigator for enrollment qualification.
* Once identified, these prospective participants will be referred to the Director of Outreach or a Good Food Rx Coordinator and/or Health Educator who will contact them to schedule an appointment to discuss the study and sign the informed consent and HIPAA Research Authorization forms if so desired.
* The prospective participants will be asked to come to the clinic to meet with study personnel in their offices for this intake. This visit is considered a research-only function that will not consume any clinical space or clinical staff time.
* If a participant decides to be in the study, in addition to signing the informed consent and HIPAA Research Authorization forms , they will be asked to sign an enrollment application, a photography release agreement consent form and complete a pre - assessment nutritional profile.
* Upon enrollment, the participant will be expected to attend bi - monthly, 30 minutes to 1 hour, nutrition education classes facilitated by UAMS East outreach staff on a variety of subjects such as meal planning, reading food labels, portion awareness, smart shopping and budgeting, as well as other topic concerning healthy eating. These bi - monthly nutrition educational classes will be present in either a group setting or individually depending on participant attendance.
* Once the participant has completed the nutrition education sessions, they will receive a free nutrition box that includes recipes using the food contents from the prepackaged box.
* Participants will be in the active study for 12 months, where the participants will attend the nutrition education classes and have their routine laboratory data collected, followed by an additional 12 months where the same data collected during the active part of the study data will be collected from the participants' electronic medical records for comparison to the active portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, 18-years old and older
* Diagnosed with a chronic health morbidity such as hypertension, elevated A1C, hyperlipidemia and/or obesity.
* A patient at UAMS East Family Medical Center in Helena, Arkansas.

Exclusion Criteria:

* Participants 17-years old and younger are excluded from The Good Food Rx program.
* Participants who are generally healthy and do not have chronic morbidities such hypertension, elevated A1C, hyperlipidemia and obesity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Blood Pressure - 3 month | 3 months
  blood pressure will be collected
Blood Pressure - 6 month | 6 months
  blood pressure will be collected
Blood Pressure - 9 month | 9 months
  blood pressure will be collected
Blood Pressure - 12 month | 12 months
  blood pressure will be collected
hemoglobin A1C - 3 month | 3 months
  routine hemoglobin A1C will be determined
hemoglobin A1C - 6 month | 6 months
  routine hemoglobin A1C will be determined
hemoglobin A1C - 9 month | 9 months
  routine hemoglobin A1C will be determined
hemoglobin A1C - 12 month | 12 months
  routine hemoglobin A1C will be determined
Total Cholesterol - 6 month | 6 month
  total cholesterol will be determined from routine clinic visits
Total Cholesterol - 12 month | 12 month
  total cholesterol will be determined from routine clinic visits
Body Weight - 3 month | 3 month
  Body weigh in lbs will be collected at routine clinic visits
Body Weight - 6 month | 6 month
  Body weigh in lbs will be collected at routine clinic visits
Body Weight - 9 month | 9 month
  Body weigh in lbs will be collected at routine clinic visits
Body Weight - 12 month | 12 month
  Body weigh in lbs will be collected at routine clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Amber K Norris, MD, Principal Investigator — UAMS
Locations (1):
- UAMS East - Helena, Helena, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided